CLINICAL TRIAL: NCT02254707
Title: A Multinational Randomised, Double-blind, Placebo Controlled Study to Evaluate the Antiviral Pharmacodynamic Effect, Safety, and Pharmacokinetics of Escalating Doses of BILB 1941 ZW Oral Solution Administered Q8H for Five Days to Patients With Chronic Hepatitis C Genotype 1 Virus Infection
Brief Title: Evaluation of the Antiviral Pharmacodynamic Effect, Safety, and Pharmacokinetics of Escalating Doses of BILB 1941 ZW to Patients With Chronic Hepatitis C Genotype 1 Virus Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1201.14
Record Dates: First submitted 2014-10-01; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (2):
- BILB 1941 ZW (Experimental): Escalating Doses
  Interventions: Drug: BILB 1941 ZW
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BILB 1941 ZW
  Arms: BILB 1941 ZW
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the antiviral effect, safety and pharmacokinetics of rising doses of 10 mg, 20 mg, 40 mg, 60 mg, 80 mg, 100 mg, 150 mg, 200 mg, 300 mg, 450 mg, 650 mg, 900 mg oral BILB 1941 ZW administered Q8H in a polyethyleneglycol 400 (PEG 400): distilled water: Tromethamine (TRIS) drinking solution for five days to patients with chronic HCV genotype 1 infection

ELIGIBILITY:
Inclusion Criteria:

1. Adult males from 18 - 65 years
2. Written informed consent consistent with ICH (International Conference on Harmonisation)/GCP (Good Clinical Practice) and local legislation given prior to any study procedures
3. Chronic HCV infection demonstrated by positive HCV IgG Antibody
4. HCV genotype 1 which has to be confirmed by central laboratory test before Visit 2
5. Liver biopsy consistent with active Hepatitis C virus (HCV) infection obtained within the last 24 months showing minimal to mild liver fibrosis and without cirrhosis (Ishak or Metavir grade <= 2)
6. HCV ribonucleic acid (RNA) load greater than 100,000 IU RNA per ml serum at screening
7. Willing to abstain from alcohol during the screening, treatment and until completion of the study (visit 11)

Exclusion Criteria:

1. Males not using an adequate form of contraception (condom, sterilisation at least 6 months post operation) in case their partner is of childbearing potential and is not using an adequate form of contraception (hormonal contraceptives, oral or injectable/implantable, intra-uterine device (IUD).
2. Any other or additional plausible cause for chronic liver disease, including the presence of other viruses known or suspected to cause hepatitis
3. Evidence of decompensated liver disease: ascites, portal hypertension or hepatic encephalopathy
4. Positive test for human immunodeficiency virus (HIV) or Hepatitis B surface (HBs) antigen at screening
5. Current alcohol or drug abuse, or history of the same, within the past twelve (12) months. All patients must abstain from alcohol from enrolment until completion of the study (visit 11).
6. Any concurrent medical illness or disease requiring treatment or concomitant medications
7. History of malignancy (except for previously cured squamous cell or basal cell carcinoma)
8. Usage of any investigational drug within thirty (30) days prior to enrolment or 5 halflives, whichever is longer; or the planned usage of an investigational drug during the course of the current study
9. Patients treated with interferon and/or ribavirin within 6 months prior to screening
10. Planned or concurrent usage of any other pharmacological therapy at screening, or during the trial period, including any antiviral therapy or vaccination
11. Known hypersensitivity to drugs or excipients
12. Patients with any one of the following laboratory values at screening:

    * Alanine transaminase (ALT) or Aspartate transaminase (AST) > 2.5 x upper limit of normal (ULN) (at screening and during the last 3 months before screening demonstrated by at least 2 further determinations)
    * Total bilirubin > 1x ULN
    * Alkaline phosphatase > 1.5x ULN
    * Prothrombin time (INR, prolonged) > 1.5
    * Platelet count < 100,000 / mm3
    * Hemoglobin < 10.5 g/dL
    * White blood cell count < 2,000 / mm3
13. Patients with any clinically significant laboratory abnormalities based on the investigator's medical assessment at screening
14. Positive urine test for drug abuse at screening
15. Patients with known Gilbert's disease
16. Prior randomisation to active treatment with BILB 1941 ZW into dose groups 3 - 9 of this trial, or previous re-treatment based on amendment 2. To support selection, centers will receive lists of the placebo patients of the previous dose levels, however, only for each center separately
17. Inability to comply with the protocol

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-07; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change in virus load (VL) | Up to day 6
  determined by IU per ml serum from baseline by > 1.0 log10 step

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Up to 14 days after first drug administration
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | Up to 14 days after first drug administration
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose) | Up to 14 days after first drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 14 days after first drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Up to 14 days after first drug administration
λz (terminal rate constant in plasma) | Up to 14 days after first drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 14 days after first drug administration
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | Up to 14 days after first drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular administration) | Up to 14 days after first drug administration
Number of patients with clinically significant changes in vital signs | Up to 14 days after first drug administration
Number of patients with clinically significant changes in body temperature | Up to 14 days after first drug administration
Number of patients with abnormal findings in electrocardiogram (ECG) | Up to 14 days after first drug administration
Number of patients with abnormal changes in clinical laboratory parameters | Up to 14 days after first drug administration
Number of patients with adverse events | Up to 14 days after first drug administration
Number of patients with abnormal findings in physical examination | Up to 14 days after first drug administration
Investigator assessed tolerability on a 4 point scale | Up to 14 days after first drug administration